CLINICAL TRIAL: NCT00456521
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Comparing the Safety and Efficacy of Naltrexone Sustained Release (SR)/Bupropion SR and Placebo in Subjects With Obesity Participating in a Behavior Modification Program
Brief Title: A Safety and Efficacy Study of Naltrexone SR/Bupropion SR and Placebo in Overweight and Obese Subjects Participating in an Intensive Behavior Modification Program
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Orexigen Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NB-302; COR-BMOD (Other: Orexigen Therapeutics, Inc.)
Record Dates: First submitted 2007-04-03; First posted 2007-04-05 (Estimated); Results first posted 2014-11-21 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Obesity; Overweight
Keywords: Obesity; Behavior Modification
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NB32 (Experimental): Naltrexone SR 32 mg/ bupropion SR 360 mg/ day with intensive group lifestyle modification counseling
  Interventions: Drug: Naltrexone SR 32 mg/ bupropion SR 360 mg/ day; Behavioral: Intensive group lifestyle modification counseling
- Placebo (Placebo Comparator): Placebo with intensive group lifestyle modification counseling
  Interventions: Drug: Placebo; Behavioral: Intensive group lifestyle modification counseling

INTERVENTIONS:
Drug: Naltrexone SR 32 mg/ bupropion SR 360 mg/ day
  Other Names: NB32
  Arms: NB32
Drug: Placebo
  Arms: Placebo
Behavioral: Intensive group lifestyle modification counseling

SUMMARY:
The purpose of this study is to determine whether a combination of naltrexone SR and bupropion SR is safe and effective in treating obesity and leads to greater weight loss when given with a group lifestyle modification program than with group lifestyle modification alone.

DETAILED DESCRIPTION:
The combination of group lifestyle modification counseling and pharmacotherapy has recently been shown to result in nearly twice the average weight loss at one year (12.1 kg) as pharmacotherapy alone (sibutramine, 5.0 kg) or lifestyle modification counseling alone (6.7 kg). Combining pharmacotherapy with a comprehensive program of diet, exercise and group lifestyle modification counseling may provide the best weight loss regimen. This study evaluated weight loss in subjects participating in such a comprehensive program who received a combination of naltrexone SR and bupropion SR, or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Female or male subjects aged 18 to 65 years (inclusive)
* Body mass index (weight [kg]/height [m²]) ≥30 and ≤45 kg/m² for subjects with uncomplicated obesity, and BMI of ≥27 and ≤45 kg/m² for subjects with controlled hypertension and/or dyslipidemia
* Non-smoker and had not used tobacco or nicotine products for at least 6 months before screening
* Normotensive (systolic ≤140 mm Hg and diastolic ≤90 mm Hg). Anti-hypertensive medications were allowed with the exception of alpha-adrenergic blockers, beta-blockers, and clonidine. Medical regimen was to be stable for at least 8 weeks.
* Low-density lipoprotein level <190 mg/dL and triglycerides level <400 mg/dL. Medications for the treatment of dyslipidemia were allowed as long as the medical regimen had been stable for at least 8 weeks.
* No clinically significant abnormality of serum albumin, blood urea nitrogen (BUN), creatinine, bilirubin, calcium and phosphorus
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) within 2.5 times upper limit of normal (ULN)
* No clinically significant abnormality of hematocrit, white blood cell (WBC) count, WBC differential, or platelets
* Fasting glucose ≤126 mg/dL and not receiving hypoglycemic agents
* No clinically significant abnormality on urinalysis
* Thyroid stimulating hormone (TSH) within 1.5 times ULN or normal triiodothyronine (T3), if TSH was below normal limits
* Female subjects of childbearing potential had a negative serum pregnancy test
* An IDS-SR score <2 on individual items: 5 (sadness), 6 (irritability), 7 (anxiety/tension), and 18 (suicidality) and an IDS-SR total score <30
* Female subjects of childbearing potential were non-lactating and agreed to continue to use effective contraception throughout the study and 30 days after discontinuation of study drug
* Completed a food diary for 6 of 7 consecutive days during screening
* Able to comply with all required study procedures and schedule
* Able to speak and read English
* Provided written informed consent

Exclusion Criteria:

* Obesity of known endocrine origin (e.g., untreated hypothyroidism, Cushing's syndrome, established polycystic ovary syndrome)
* Serious medical condition (including but not limited to renal or hepatic insufficiency; congestive heart failure, angina pectoris, myocardial infarction, stroke, claudication, or acute limb ischemia; history of malignancy with exception of non-melanoma skin cancer or surgically cured cervical cancer)
* Serious psychiatric illness (e.g., lifetime history of bipolar disorder, schizophrenia or other psychosis, bulimia, and anorexia nervosa; current serious personality disorder, e.g., borderline; severe major depressive disorder, recent [previous 6 months] suicide attempt or current active suicidal ideation, recent hospitalization due to psychiatric illness)
* Response to the bipolar disorder questions that indicated the presence of bipolar disorder.
* Required medications for the treatment of a psychiatric disorder (with the exception of short-term insomnia) within the previous 6 months
* History of drug or alcohol abuse or dependence within 1 year
* Type I or Type II diabetes mellitus
* Baseline ECG with a corrected QT (QTc) interval (using Bazett's formula >450 millisecond (msec) [males] and >470 msec [females]) or the presence of any clinically significant cardiac abnormalities, including but not limited to patterns consistent with myocardial ischemia, electrolyte abnormalities, or atrial or ventricular dysrhythmia or significant conduction abnormalities
* Received excluded concomitant medications: any psychotropic agents (including antipsychotic, antidepressant, anxiolytic, mood stabilizer or anticonvulsant agents) with the exception of low-dose benzodiazepine or hypnotic agents for the treatment of insomnia; any anorectic or weight loss agents; any over-the-counter dietary supplements with psychoactive, appetite or weight effects; alpha-adrenergic blockers; beta-blockers; clonidine; coumadin; theophylline; cimetidine; oral corticosteroids; topiramate, Depo-Provera®; smoking cessation agents; regular use of opioid or opioid-like analgesics
* History of surgical or device (e.g., lap band) intervention for obesity
* History of seizures of any etiology, or of predisposition to seizures (e.g., history of cerebrovascular accident, head trauma with >5 minutes loss of consciousness, concussion symptoms lasting >15 minutes, brain surgery, skull fracture, subdural hematoma, or febrile seizures)
* History of treatment with bupropion or naltrexone within the preceding 12 months
* History of hypersensitivity or intolerance to bupropion or naltrexone
* Used drugs, herbs, or dietary supplements believed to significantly affect body weight or participated in a weight loss management program within one month prior to baseline
* Loss or gained >4.0 kilograms within the previous 3 months
* Females who were pregnant or breast-feeding or planning to become pregnant during the study period or within 30 days of discontinuing study drug
* Planned surgical procedure that could impact the conduct of the study
* Received any investigational drug or used an experimental device or procedure within the previous 30 days
* Participated in any previous clinical trial conducted by Orexigen
* Had any condition that in the opinion of the investigator made the subject unsuitable for inclusion into the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 793 (Actual)
Dates: Start 2007-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of California, San Diego: Dept of Family & Preventive Medicine, La Jolla, California
  - Center for Human Nutrition, University of Colorado Health Services Center, Denver, Colorado
  - Univ. of Florida, College of Public Health, and Health Professions, Gainesville, Florida
  - Washington Univ. Center for Human Nutrition, St Louis, Missouri
  - New York Obesity Research Center, St. Luke's-Roosevelt Hospital Center, New York, New York
  - Center for Weight and Eating Disorders, School of Med., University of Penn., Philadelphia, Pennsylvania
  - Center for Obesity Research and Education, Temple University, Philadelphia, Pennsylvania
  - Medical University of S. Carolina Weight Management Center, Charleston, South Carolina
  - Behavioral Medicine Research Center, Houston, Texas

REFERENCES:
- [Result] Wadden TA, Foreyt JP, Foster GD, Hill JO, Klein S, O'Neil PM, Perri MG, Pi-Sunyer FX, Rock CL, Erickson JS, Maier HN, Kim DD, Dunayevich E. Weight loss with naltrexone SR/bupropion SR combination therapy as an adjunct to behavior modification: the COR-BMOD trial. Obesity (Silver Spring). 2011 Jan;19(1):110-20. doi: 10.1038/oby.2010.147. Epub 2010 Jun 17. PMID 20559296

RESULTS

PARTICIPANT FLOW:
Groups:
- NB32: Naltrexone SR 32 mg/ bupropion SR 360 mg/ day
- Placebo: Placebo
Period: Overall Study
Arm/Group | NB32 | Placebo
Started | 591 | 202
Completed | 342 | 118
Not Completed | 249 | 84
Not completed — Adverse Event | 150 | 25
Not completed — Withdrawal by Subject | 43 | 24
Not completed — Lost to Follow-up | 22 | 17
Not completed — Lack of Efficacy | 3 | 6
Not completed — Protocol Violation | 4 | 0
Not completed — Pregnancy | 1 | 1
Not completed — Drug non-compliance, moved, other | 26 | 11

BASELINE CHARACTERISTICS:
Population: All randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | NB32 | Placebo | Total
Number analyzed (Participants) | 591 | 202 | 793
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.89 (10.42) | 45.59 (11.35) | 45.82 (10.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 528 | 185 | 713
  Male | 63 | 17 | 80
Race/Ethnicity, Customized [Number; unit: participants]
  White | 405 | 149 | 554
  Black or African American | 145 | 44 | 189
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  American Indian or Alaska Native | 7 | 1 | 8
  Other | 27 | 6 | 33
Weight [Mean (Standard Deviation); unit: kg] | 100.16 (15.42) | 101.88 (14.96) | 100.60 (15.31)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 36.34 (4.16) | 36.96 (4.18) | 36.50 (4.17)

OUTCOME MEASURES:

1. Primary Outcome: Co-primary: Body Weight- Mean Percent Change
Time Frame: Baseline, 56 weeks
Population: Modified ITT (Full Analysis Set): Included all subjects who were randomized, had a baseline weight measurement, and had at least one post-baseline weight measurement while on study drug. Missing data were imputed with the LOCF method.
Measure: Least Squares Mean (Standard Error); unit: percentage of body weight
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 482 | 193
percentage of body weight | -9.29 (0.40) | -5.08 (0.60)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -4.21, 95% CI [-5.56 to -2.86]

2. Primary Outcome: Co-primary: Body Weight- Proportion of Subjects With ≥5% Decrease
Time Frame: Baseline, 56 weeks
Population: Modified ITT: Included all subjects who were randomized, had a baseline weight measurement, and had at least one post-baseline weight measurement while on study drug. Missing data were imputed with the LOCF method.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 482 | 193
percentage of participants | 66.39 [62.17 to 70.61] | 42.49 [35.51 to 49.46]
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.89, 95% CI [2.02 to 4.13]

3. Secondary Outcome: Body Weight- Proportion of Subjects With ≥10% Decrease
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 482 | 193
percentage of participants | 41.49 [37.10 to 45.89] | 20.21 [14.54 to 25.87]
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.92, 95% CI 2-sided [1.95 to 4.37]

4. Secondary Outcome: Change in Waist Circumference
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 391 | 141
cm | -9.98 (0.48) | -6.77 (0.75)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -3.21, 95% CI 2-sided [-4.82 to -1.60]

5. Secondary Outcome: Change in Fasting Triglycerides Levels, Using Log-transformed Data
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 392 | 144
percent change | -16.62 [-19.66 to -13.47] | -8.51 [-13.67 to -3.03]
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p = 0.004, ANCOVA; Mean Difference (Net) = -8.11

6. Secondary Outcome: Change in Fasting Insulin Levels, Using Log-transformed Data
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 386 | 144
percent change | -27.98 [-32.36 to -23.31] | -15.45 [-23.29 to -6.81]
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p = 0.003, ANCOVA; Mean Difference (Net) = -12.53

7. Secondary Outcome: Change in Fasting HDL Cholesterol Levels
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 392 | 144
mg/dL | 4.10 (0.51) | 0.87 (0.80)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = 3.23, 95% CI 2-sided [1.52 to 4.95]

8. Secondary Outcome: Change in IWQOL-Lite Total Scores
Description: IWQOL-Lite= Impact of Weight on Quality of Life-Lite Questionnaire Total score is based on a scale from 0 to 100, with 0 representing the poorest and 100 the best quality of life and where a score of 71-79 indicates moderate impairment
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 448 | 178
units on a scale | 13.43 (0.56) | 10.29 (0.86)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA; Mean Difference (Net) = 3.14, 95% CI 2-sided [1.23 to 5.04]

9. Secondary Outcome: Change in HOMA-IR Levels, Using Log-transformed Data
Description: HOMA-IR= Homeostasis Model Assessment-Insulin Resistance
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 385 | 143
percent change | -29.93 [-34.59 to -24.93] | -16.56 [-25.02 to -7.14]
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p = 0.003, ANCOVA; Mean Difference (Net) = -13.37

10. Secondary Outcome: Change in High-sensitivity C Reactive Protein (Hs-CRP) Levels, Using Log-transformed Data
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 386 | 143
percent change | -25.87 [-32.58 to -18.49] | -16.89 [-28.31 to -3.66]
Statistical Analysis 1: Comparison: NB32 vs Placebo; Test type: Superiority or Other; p = 0.165, ANCOVA; Mean Difference (Net) = -8.98

11. Secondary Outcome: Change in Fasting Blood Glucose Levels
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 393 | 144
mg/dL | -2.36 (0.62) | -1.08 (0.96)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = -1.28, 95% CI 2-sided [-3.34 to 0.79]

12. Secondary Outcome: Change in Fasting LDL Cholesterol
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 392 | 143
mg/dL | 5.43 (1.36) | 8.13 (2.13)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = -2.70, 95% CI 2-sided [-7.26 to 1.86]

13. Secondary Outcome: Change in Systolic Blood Pressure
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 482 | 193
mmHg | -1.32 (0.47) | -3.87 (0.71)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = 2.55, 95% CI 2-sided [0.97 to 4.14]

14. Secondary Outcome: Change in Diastolic Blood Pressure
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 482 | 193
mmHg | -1.41 (0.33) | -2.78 (0.50)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = 1.37, 95% CI 2-sided [0.25 to 2.49]

15. Secondary Outcome: Change in IDS-SR Total Scores
Description: IDS-SR= Inventory of Depressive Symptoms-Subject Rated IDS-SR total score is based on 30 items. The total score can range from 0-84, with 0 being no depressive symptoms and 84 being very severe depressive symptoms. A total score ≤ 13 indicates no depression.
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 482 | 193
units on a scale | 0.09 (0.23) | -0.00 (0.35)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = 0.09, 95% CI 2-sided [-0.70 to 0.87]

16. Secondary Outcome: Change in Food Craving Inventory Sweets Subscale Scores
Description: The Food Craving Inventory is a 33-item self-report measure designed to assess specific food cravings and is organized into 4 subscales (high fats, sweets, carbohydrates/starches, and fast-food fats). A craving was defined as an intense desire to consume a particular food (or food type) that was difficult to resist over the past month. Subjects rated their frequency of cravings for each of the 33 items using a 5-point scale, where 1=never, 2=rarely, 3=sometimes, 4=often, and 5=always. The sweets subscale consisted of 8 items and the score ranges from 8 (better outcome) to 40 (worse outcome).
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 448 | 180
units on a scale | -2.54 (0.22) | -2.43 (0.33)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.85 to 0.63]

17. Secondary Outcome: Change in Food Craving Inventory Carbohydrates Subscale Scores
Description: The Food Craving Inventory is a 33-item self-report measure designed to assess specific food cravings and is organized into 4 subscales (high fats, sweets, carbohydrates/starches, and fast-food fats). A craving was defined as an intense desire to consume a particular food (or food type) that was difficult to resist over the past month. Subjects rated their frequency of cravings for each of the 33 items using a 5-point scale, where 1=never, 2=rarely, 3=sometimes, 4=often, and 5=always. The carbohydrates subscale consisted of 8 items and the score ranges from 8 (better outcome) to 40 (worse outcome).
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- NB32: Naltrexone SR 32 mg/ bupropion SR 360 mg/ day with intensive group behavioral lifestyle modification counseling
  naltrexone SR/bupropion SR combination
  Intensive group lifestyle modification counseling: Group lifestyle modification counseling
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 448 | 180
units on a scale | -2.06 (0.20) | -1.97 (0.31)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.78 to 0.60]

18. Secondary Outcome: Change in Question 19 From 21-Item COE (Control of Eating) Questionnaire
Description: Question 19: Generally, how difficult has it been to control your eating? Scoring: 0=not at all difficult; 100=extremely difficult
Time Frame: Baseline, 56 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NB32 | Placebo
Number analyzed (Participants) | 436 | 178
units on a scale | -13.75 (1.17) | -8.46 (1.75)
Statistical Analysis 1: Comparison: NB32 vs Placebo; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Test type: Superiority or Other; Due to pre-specified hypothesis testing design, no formal statistical inference testing was performed; Mean Difference (Net) = -5.29, 95% CI 2-sided [-9.16 to -1.42]

ADVERSE EVENTS:
Time Frame: Baseline, 56 weeks
Description: The safety analysis set includes all randomized subjects who took study drug and were assessed by investigator after their first dose, whether or not they discontinue the study.Treatment-emergent adverse events were defined as events that started or worsened in the double-blind treatment phase after the first dose and before 30 days post last dose.
Arm/Group | NB32 | Placebo
Serious Adverse Events (participants affected / at risk) | 22/584 | 1/200
Other Adverse Events (participants affected / at risk) | 465/584 | 132/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NB32 (N=584) | Placebo (N=200)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Epiploic appendagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 4 (4) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis acute (Infections and infestations) | 1 (1) | 0 (0)
Bursitis infective (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NB32 (N=584) | Placebo (N=200)
Tinnitus (Ear and labyrinth disorders) | 31 (33) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 32 (33) | 3 (4)
Constipation (Gastrointestinal disorders) | 141 (157) | 28 (32)
Diarrhoea (Gastrointestinal disorders) | 43 (45) | 15 (16)
Dry mouth (Gastrointestinal disorders) | 47 (48) | 6 (6)
Nausea (Gastrointestinal disorders) | 199 (228) | 21 (21)
Vomiting (Gastrointestinal disorders) | 64 (76) | 13 (13)
Fatigue (General disorders) | 31 (35) | 13 (13)
Nasopharyngitis (Infections and infestations) | 36 (41) | 15 (18)
Upper respiratory tract infection (Infections and infestations) | 38 (40) | 18 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 28 (33) | 12 (12)
Dizziness (Nervous system disorders) | 85 (96) | 9 (10)
Headache (Nervous system disorders) | 139 (167) | 35 (42)
Tremor (Nervous system disorders) | 34 (41) | 2 (2)
Anxiety (Psychiatric disorders) | 30 (34) | 7 (7)
Insomnia (Psychiatric disorders) | 51 (51) | 12 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 28 (35) | 15 (18)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 20 (23) | 10 (12)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 29 (36) | 17 (19)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 18 (20) | 13 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If not already published by Sponsor as part of a multi-center publication, 18 months after conclusion of the study at all study centers, PI may publish the results for PI's study center individually. Prior to such publication, PI must provide Sponsor with at least 60 days to review and comment on the proposed publication. The review period may be extended by an additional 30 days upon request. Sponsor may delay publication for up to an additional 6 month period to file for patent protection.